CLINICAL TRIAL: NCT01005030
Title: Evaluation of Blood Biospectroscopy as a Novel Diagnostic Test for Idiopathic Parkinson Disease
Brief Title: Spectroscopy in Parkinson Disease
Acronym: SPIN-PD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Molecular Biometrics, Inc. (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Bruce J. Goldstein / Vice President, Operations, Molecular Biometrics, Inc.
Other Study IDs: MB_PD001
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; blood; plasma; metabolomics; spectroscopy; oxidative stress.
MeSH Terms: conditions — Parkinson Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma, cell free
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PostCEPT Subjects: Subjects with current Parkinson Disease Diagnosis currently enrolled in PostCEPT study
  Interventions: Other: Blood draw
- Control Subjects: Non-blood relatives of PostCEPT Subjects matched for age and other demographics
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — Blood draw, two tubes, used for isolation of cell-free blood plasma

SUMMARY:
The primary objective of the study is to determine the utility of blood plasma infrared spectroscopy (biospectroscopy) in distinguishing subjects with idiopathic Parkinson's disease from healthy controls.

DETAILED DESCRIPTION:
Oxidative stress has been implicated as a factor in the pathogenesis of Parkinson's disease (PD). The overall goal of this proposal is to use a novel metabolomics platform, based on near infrared biospectroscopy, to detect oxidatively modified blood plasma constituents. These spectral findings can be used to model the degree of oxidative stress with a modeled "stress index" that may distinguish PD cases from healthy elderly controls.

ELIGIBILITY:
Inclusion Criteria:

PD Subjects:

1. PostCEPT subjects with a diagnosis of PD based on UK Brain Bank criteria.
2. Willing and able to provide informed consent.

Healthy Controls:

1. No current diagnosis or known history of a neurological disease/disorder.
2. Non-blood relative of a patient or subject at the site who has diagnosis of PD (may include healthy controls from the PROBE study).
3. No first degree relatives with diagnosis of PD
4. MoCA score > 26.
5. Age > 45.
6. Willing and able to provide informed consent.

Min Age: 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's subjects: from pool of subjects currently enrolled in PostCEPT study Control subjects: general population
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of the study is the correct classification of cases of PD and controls. This will be quantified as sensitivity and specificity. | Baseline and annually for two years

SECONDARY OUTCOMES:
Determine impact of disease stage, age, gender, medications, cognitive scores, other laboratory measures (e.g. alpha-synuclein) and other clinical/demographic variables on plasma biospectra. | Baseline and annually for two years
Correlate plasma biospectra with dopamine transporter neuroimaging data. | Baseline and annually for two years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Ravina, MD, Principal Investigator — University of Rochester; Anthony E Lang, MD, Principal Investigator — University of Toronto
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Background] Burns DH, Rosendahl S, Bandilla D, Maes OC, Chertkow HM, Schipper HM. Near-infrared spectroscopy of blood plasma for diagnosis of sporadic Alzheimer's disease. J Alzheimers Dis. 2009;17(2):391-7. doi: 10.3233/JAD-2009-1053. PMID 19363272
- [Background] Schipper HM, Kwok CS, Rosendahl SM, Bandilla D, Maes O, Melmed C, Rabinovitch D, Burns DH. Spectroscopy of human plasma for diagnosis of idiopathic Parkinson's disease. Biomark Med. 2008 Jun;2(3):229-38. doi: 10.2217/17520363.2.3.229. PMID 20477412
- See also: The Parkinson Study Group (PSG) is a non-profit, cooperative group of Parkinson's disease experts from medical centers in the United States and Canada who are dedicated to improving treatment for persons affected by Parkinson's disease. — http://www.parkinson-study-group.org